CLINICAL TRIAL: NCT07375563
Title: Chemoimmunotherapy Combined With Autologous NK Cell Therapy for the Treatment of Pediatric Patients With Refractory and Relapsed High-Risk Neuroblastoma and Ganglioneuroblastoma
Brief Title: Chemoimmunotherapy Combined With Autologous NK Cell Therapy for Pediatric Patients With Refractory and Relapsed High-Risk Neuroblastoma and Ganglioneuroblastoma
Acronym: NB-NK-2026
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCHPOI- 2025-10
Record Dates: First submitted 2026-01-15; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Neuroblastoma (NB); Ganglioneuroblastoma
Keywords: Refractory/relapsed neuroblastoma; ganglioneuroblastoma; children; autologous NK cells; chemoimmunotherapy; dinutuximab beta
MeSH Terms: conditions — Neuroblastoma; Ganglioneuroblastoma | interventions — dinutuximab; Temozolomide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm А: patients with a refractory disease (Experimental): Patients who meet the inclusion criteria will undergo an intensified induction phase within the framework of this clinical trial protocol, while the preceding induction phase and subsequent consolidation and post-consolidation phases will be performed outside of this protocol in accordance with the current clinical practice. As part of the intensified induction, a procedure for the collection of mononuclear cells for the cultivation and expansion of the autologous NK cell product (Day -1) is planned, followed by one course of chemotherapy according to the IT regimen (irinotecan + temozolomide) and four courses of chemoimmunotherapy in combination with autologous NK cell therapy according to the DIT regimen (irinotecan + temozolomide + dinutuximab beta + NK-cell product)
  Interventions: Combination Product: Dinutuximab beta, temozolomide, irinotecan, autologous NK cell; Combination Product: irinotecan, temozolomide, dinutuximab beta, NK-cell product
- Arm B: patients with relapsed/ progression disease (Experimental): Patients who meet the inclusion criteria will undergo peripheral blood collection with subsequent isolation of mononuclear cells for cultivation and expansion of an autologous NK cell product (Day -1), followed by administration of the first course of chemotherapy according to the IT regimen (irinotecan + temozolomide) and five courses of chemoimmunotherapy in combination with autologous NK cell therapy according to the DIT regimen (irinotecan + temozolomide + dinutuximab beta + autologous NK cell product)
  Interventions: Combination Product: Dinutuximab beta, temozolomide, irinotecan, autologous NK cell; Combination Product: irinotecan, temozolomide, dinutuximab beta, NK-cell product

INTERVENTIONS:
Combination Product: Dinutuximab beta, temozolomide, irinotecan, autologous NK cell — As part of the intensified induction, a procedure for the collection of mononuclear cells for the cultivation and expansion of the autologous NK cell product (Day -1) is planned, followed by one course of chemotherapy according to the IT regimen (irinotecan + temozolomide) and four courses of chemoimmunotherapy in combination with autologous NK cell therapy according to the DIT regimen (irinotecan + temozolomide + dinutuximab beta + NK-cell product), with an inter-cycle interval of 21 days. Transfusion of the autologous NK cell product will be performed on Day 7 of each DIT course.
Combination Product: irinotecan, temozolomide, dinutuximab beta, NK-cell product — Patients who meet the inclusion criteria will undergo an intensified induction phase within the framework of this clinical trial protocol, while the preceding induction phase and subsequent consolidation and post-consolidation phases will be performed outside of this protocol in accordance with the current clinical practice. As part of the intensified induction, a procedure for the collection of mononuclear cells for the cultivation and expansion of the autologous NK cell product (Day -1) is planned, followed by one course of chemotherapy according to the IT regimen (irinotecan + temozolomide) and four courses of chemoimmunotherapy in combination with autologous NK cell therapy according to the DIT regimen (irinotecan + temozolomide + dinutuximab beta + NK-cell product)

SUMMARY:
Neuroblastoma (NB) is a malignant neoplasm of the sympathetic nervous system, occurring in 1 in 8,000 live births, accounting for 6-10% of all childhood malignant neoplasms and responsible for 12-15% of mortality -, making it the most common and life-threatening extracranial tumor in childhood.

Patients with stage 4 high-risk NB is the subgroup with the poorest prognosis. Within this group, two subgroups with an extremely unfavorable disease course are distinguished: patients with a poor response to the induction phase of therapy (refractory disease) and patients with relapsed or progressive disease.

Nowadays, 10-15% of patients show a poor end-induction response, whereas achieving a good end-induction response associated with better long-term survival. Improvement of the response to induction therapy may contribute to better treatment outcomes in newly diagnosed high-risk NB patients and can be achieved by intensification of the induction phase to decrease the number of patients with refractory disease. Also intensification of the second-line therapy may contribute to better responses in patients with relapsed and progressive disease.

Protocol aimed to overcome heterogeneous tumor drug resistance through the synergistic interaction of cytostatic and immunobiological agents in combination with NK cell therapy.

This approach combines cytotoxic agents with anti-GD2 monoclonal antibodies (mAb) to enhance antitumor activity. Cultured, ex vivo-activated autologous NK cells are infused to compensate for effector cell depletion during therapy and to augment antibody-dependent cellular cytotoxicity (ADCC), potentially improving clinical outcomes.

This comprehensive approach opens novel prospects for enhancing treatment efficacy in patients with refractory and relapsed high-risk NB.

The expected outcomes of this protocol include a significant increase in therapeutic efficacy indicators - objective response rate (ORR), overall survival (OS), progression-free survival (PFS) and relapse-free survival (RFS), as well as in patient quality of life.

DETAILED DESCRIPTION:
The study design evaluates a therapeutic interventionin two independent groups:

1. Arm А: patients with a refractory disease
2. Arm B: patients with relapsed/ progression disease

Intervention plan for patients with a refractory NB (arm A):

Patients who meet the inclusion criteria will undergo an intensified induction phase within the framework of this clinical trial protocol, while the preceding induction phase and subsequent consolidation and post-consolidation phases will be performed outside of this protocol in accordance with the current clinical practice. As part of the intensified induction, a procedure for the collection of mononuclear cells for the cultivation and expansion of the autologous NK cell product (Day -1) is planned, followed by one course of chemotherapy according to the IT regimen (irinotecan + temozolomide) and four courses of chemoimmunotherapy in combination with autologous NK cell therapy according to the DIT regimen (irinotecan + temozolomide + dinutuximab beta + NK-cell product), with an inter-cycle interval of 21 days. Transfusion of the autologous NK cell product will be performed on Day 7 of each DIT course.

Intervention plan for patients with relapsed/progression (arm В):

Patients who meet the inclusion criteria will undergo peripheral blood collection with subsequent isolation of mononuclear cells for cultivation and expansion of an autologous NK cell product (Day -1), followed by administration of the first course of chemotherapy according to the IT regimen (irinotecan + temozolomide) and five courses of chemoimmunotherapy in combination with autologous NK cell therapy according to the DIT regimen (irinotecan + temozolomide + dinutuximab beta + autologous NK cell product) with a 21-day inter-cycle interval within the framework of this clinical trial protocol. Subsequent phases of therapy (including delayed surgery and external beam radiotherapy) will be carried out after completion of the chemoimmunotherapy in combination with autologous NK cell therapy, outside the present protocol, in accordance with current clinical practice. Transfusion of the autologous NK cell product will be performed on Day 7 of each DIT course.

ELIGIBILITY:
Inclusion Criteria:

* Signed voluntary informed consent to participate in the clinical trial
* Histologically verified diagnosis of neuroblastoma or ganglioneuroblastoma
* Patients stratified to the high-risk group according to the criteria of the German Society of Pediatric Oncology and Hematology (GPOH) - NB 2004, aged from 18 months to 18 years, and meeting the following conditions:

  1. Arm A: Refractory disease - patients who have completed the induction phase of therapy (6 cycles of N5/N6) with a poor response to therapy (MR, SD), with the exception of PD
  2. Arm В: Relapsed/progressive disease - patients who develop any new tumor lesions (after having previously achieved СR), or any new tumor lesion; an increase of >25% in any previously existing measurable lesion; or newly detected bone marrow involvement by NB cells in cases where the bone marrow had previously been free of involvement
* Performance status ≥ 70% (Lansky or Karnofsky scale) at the time of determining the indication for chemoimmunotherapy combined with NK cell therapy.
* Expected life expectancy ≥ 12 weeks.
* No signs of drug-induced neuropathy or neuropathic pain.
* Adequate liver function: alanine aminotransferase (ALT) / aspartate aminotransferase (AST) activity < 5 × upper limit of normal (ULN).
* Adequate renal function: creatinine clearance or glomerular filtration rate (GFR) > 60 mL/min/1.73 m².
* Coagulation parameters: prothrombin index (PTI) 70-120%; activated partial thromboplastin time (APTT) < 36 seconds.
* No clinical signs of heart failure; left ventricular ejection fraction (LVEF) ≥ 55%.
* Adequate respiratory function (oxygen saturation by pulse oximetry > 94% on room air, no dyspnea at rest), and no pathological findings on chest X-ray.
* Completion of comprehensive assessment to evaluate the extent of the tumor process.

Exclusion Criteria:

* Lack of a signed voluntary informed consent form for participation in the clinical study.
* Absence of comprehensive pre-treatment assessment results at the time of initiation of specific therapy.
* Patients with NBL or ganglioneuroblastoma stratified to low or intermediate-risk group
* Good response (PR, VGPR, CR) or PD at the end of the induction phase of therapy (applicable only to patients receiving therapy within the framework of the intensified induction phase).
* Progressive or relapsed disease with central nervous system involvement and/or leptomeningeal involvement.
* History of acute intolerance reactions to the main chemotherapeutic and immunobiological agents and supportive care drugs used in this clinical trial protocol.
* Presence of complications of the underlying disease and comorbidities that preclude treatment within this protocol, including severe type I hypersensitivity reactions in the medical history.
* Requirement for concomitant medications with known cross pharmacodynamic interactions with the drugs used in this clinical trial protocol.
* Presence of ultrasonographic signs of heart failure (LVEF ≤ 55%), clinical and laboratory signs of chronic kidney disease of stage ≥ III, or kidney injury of grade I, F or L according to the standardized RIFLE criteria for acute kidney injury (an acronym for "risk, injury, failure, loss, end-stage").
* Pregnancy, due to the high teratogenicity and toxicity of the drugs used in this clinical trial protocol. Female patients of childbearing potential are required to undergo pregnancy testing.
* Mental illness of the patient or legal guardians that makes it impossible to understand the nature of the study and compromises adherence to medical prescriptions and sanitary-hygienic requirements.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2028-11-19 (Estimated)

PRIMARY OUTCOMES:
Tolerability and toxicity of chemoimmunotherapy in combination with NK cell therapy. | immediately after completion of courses of chemoimmunotherapy in combination with NK cell therapy.
  (Proportion of patients receiving at least 80% of the planned doses without grade ≥ 3 adverse immunological reactions (ADRs) related to the NK cell product, assessed acc

SECONDARY OUTCOMES:
ORR after completion of chemoimmunotherapy courses in combination with NK cell therapy. | immediately after completion of courses of chemoimmunotherapy in combination with
  (The proportion of patients with a good response (CR, VGPR and PR) to therapy, assessed in accordance with the International Response Criteria for Patients with NB)
ORR after completion of study therapy. | immediately after completion of study therapy.
  (The proportion of patients who achieved a good response (CR, VGPR and PR) to therapy, assessed in accordance with the International Response Criteria for Patients with NB)).
OS and EFS at 1 year, 3 years, and 5 years after completion of study therapy. | 1 year, 3 years, and 5 years from the date of diagnosis.
  For patients with refractory disease: The proportion of surviving patients, regardless of disease status (for OS) and the proportion of patients without adverse events, such as relapse, progression or death (for EFS)).
OS, PFS, and RFS at 1 and 3 years after completion of the study therapy. | are 1, 3, and 5 years from the date of diagnosis (for OS) or from the date of documented progression/relapse (for PFS and RFS)).
  For patients with progression/relapsed disease: The proportion of surviving patients from the time of diagnosis, regardless of disease status (for OS); the proportion of patients without disease relapse (for RFS) or disease progression (for PFS) from the time of the relapse or progression).

CONTACTS AND LOCATIONS:
Overall Officials: Tatyana V Shamanskaya, MD, PHD, Study Director — Dmitry Rogachev National Medical Research Center of Pediatric Hematology, Oncology and Immunology
Locations (1):
- National medical research center of pediatric haematology, oncology and immulogy named after Dmytriy Rogachyov, Moscow, 117198, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No